CLINICAL TRIAL: NCT00102531
Title: Phase Ib/IIa Study of SLIT Cisplatin by Inhalation in the Treatment of Patients Wtih Relapsed/Progressive Osteosarcoma Metastatic to the Lung
Brief Title: Inhalation SLIT Cisplatin (Liposomal) for the Treatment of Osteosarcoma Metastatic to the Lung
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR02-2421
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Osteosarcoma Metastatic
Keywords: Osteosarcoma; relapsed; progressive; metastatic; lung
MeSH Terms: conditions — Osteosarcoma; Recurrence; Neoplasm Metastasis | interventions — SPI-77, liposomal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cisplatin liposomal 24 mg/m2 (Experimental): Inhaled liposomal cisplatin was administered over 1 day in a 14-day treatment cycle by inhalation for a maximum of 6 cycles.
  Interventions: Drug: Cisplatin liposomal
- Cisplatin liposomal 36 mg/m2 (Experimental): The study allowed for a dose escalation of liposomal cisplatin to 36 mg/m2 if no adverse events of Grade 3 or higher occurred after at least 3 cycles of drug administration at 24 mg/m2
  Interventions: Drug: Cisplatin liposomal

INTERVENTIONS:
Drug: Cisplatin liposomal
  Other Names: SLIT Cisplatin

SUMMARY:
Phase Ib/IIa open label safety and efficacy study designed to determine the maximum tolerated dose of inhaled cisplatin liposomal (SLIT cisplatin) administered every 14 days to patients with relapsed/progressive osteosarcoma metastatic to the lung.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, Progressive or recurrent high grade osteosarcoma metastatic to the lung
* Patients with histologically proven, fully malignant high-grade osteosarcoma of bone
* Measureable pulmonary metastases
* Less than grade 3 neuropathies, insignificant decreases in cardiac or auditory function
* ECOG performance status of 0, 1 or 2
* FEV1 of 50% or greater of predicted value
* FEV1/FVC ratio of 65% or greater
* Serum creatinine of ≤ 1.5 mg/dl
* Total bilirubin ≤ 1.5mg/dl and SGOT or SGPT < 2.5 times upper normal limit
* ANC of ≥ 1,000/mm3 and platelet count of ≥ 100,000/mm3

Exclusion Criteria:

* Grade 3 or higher painful neuropathy persisting after a prior platinum containing regimen
* Patients who are pregnant or are of childbearing potential and not using methods to avoid pregnancy
* Concurrent systemic chemotherapy
* Greater than Grade 2 pulmonary toxicity
* Pulmonary atelectasis
* Reactive airway disease which has resulted in hospitalization within the last year or which requires daily treatment with bronchodilator therapy
* Concurrent serious infections
* Unstable or serious concurrent medical condition
* Recent major surgery or thoracic radiation therapy or chemotherapy
* Significant pulmonary fibrosis secondary to prior radiation
* Major ventilatory distribution abnormalities
* Osteosarcoma secondary to radiation or premalignant conditions
* History of prior malignancy
* Low grade osteosarcoma, parosteal or periosteal sarcoma

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-01-12 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renu Gupta, MD, Study Chair — Transave Inc.; Richard Gorlick, MD, Principal Investigator — The Albert Einstein College of Medicine Montefiore Medical Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Albert Einstein College of Medicine Montefiore Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chou AJ, Gupta R, Bell MD, Riewe KO, Meyers PA, Gorlick R. Inhaled lipid cisplatin (ILC) in the treatment of patients with relapsed/progressive osteosarcoma metastatic to the lung. Pediatr Blood Cancer. 2013 Apr;60(4):580-6. doi: 10.1002/pbc.24438. Epub 2012 Dec 19. PMID 23255417
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23255417

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin Liposomal 24 mg/m2: Inhaled liposomal cisplatin was administered over 1 day in a 14-day treatment cycle by inhalation for a maximum of 6 cycles.
  Cisplatin liposomal
- Cisplatin Liposomal 36 mg/m2: The study allowed for a dose escalation of liposomal cisplatin to 36 mg/m2 if no adverse events of Grade 3 or higher occurred after at least 3 cycles of drug administration at 24 mg/m2
  Cisplatin liposomal
Period: Overall Study
Arm/Group | Cisplatin Liposomal 24 mg/m2 | Cisplatin Liposomal 36 mg/m2
Started | 7 | 12
Completed | 2 | 1
Not Completed | 5 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Disease Progression | 5 | 9
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin Liposomal 24 mg/m2 | Cisplatin Liposomal 36 mg/m2 | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (4.8) | 17.8 (2.3) | 18.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 2 | 10 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 9 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: The Study Medication Was to be Considered Effective if the Population Response Rate Was Found to be Greater Than 20% and Individuals Who Demonstrated a CR or PR or Whose Tumours Demonstrated a Grade 3 or 4 Histologic Response at the Time of Surgery.
Time Frame: 4 to 48 weeks
Measure: Number; unit: participants
Groups:
- Cisplatin Liposomal 24 mg/m2: Inhaled liposomal cisplatin was administered over 1 day in a 14-day treatment cycle by inhalation
Arm/Group | Cisplatin Liposomal 24 mg/m2 | Cisplatin Liposomal 36 mg/m2
Number analyzed (Participants) | 7 | 12
participants
  CR/PR | 2 | 2
  Histological response | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs were followed until resolution until 30 days post last dose.
Arm/Group | Cisplatin Liposomal 24 mg/m2 | Cisplatin Liposomal 36 mg/m2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/12
Other Adverse Events (participants affected / at risk) | 4/7 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin Liposomal 24 mg/m2 (N=7) | Cisplatin Liposomal 36 mg/m2 (N=12)
Vomiting (Gastrointestinal disorders) | 1 | 0
pyrexia (General disorders) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin Liposomal 24 mg/m2 (N=7) | Cisplatin Liposomal 36 mg/m2 (N=12)
Gastrointestinal Disorders (Gastrointestinal disorders) | 2 | 4
General Disorders and Admin Site Conditions (General disorders) | 1 | 2
Respiratory, Thoracic and Mediastinal Disorders (Reproductive system and breast disorders) | 3 | 7
Nervous System Disorders (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No